CLINICAL TRIAL: NCT00994344
Title: Randomised and Prospective Clinical Study to Evaluate the Efficacy and Safety of Lopinavir/Ritonavir Monotherapy Versus Darunavir/Ritonavir Monotherapies as Simplification Switching Strategies of PI/NNRTI-Triple Therapy Based-Regimens
Brief Title: Clinical Study to Evaluate the Efficacy and Safety of Lopinavir/Ritonavir Monotherapy Versus Darunavir/Ritonavir Monotherapies as Simplification Switching Strategies of PI/NNRTI-Triple Therapy Based-Regimens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Sílvia Gel, Dr. Bonaventura Clotet, Germans Trias i Pujol Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LOPIDAR
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: HIV Infections
Keywords: Darunavir; Lopinavir; Monotherapy; Antiretroviral simplification strategy; HIV; Treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Darunavir; Ritonavir; Lopinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Darunavir/ritonavir (Experimental): to switch from the triple therapy based regimens to Darunavir/ritonavir
  Interventions: Drug: Darunavir/ritonavir
- Lopinavir/ritonavir (Active Comparator): to switch from the triple therapy based regimens to Lopinavir/ritonavir
  Interventions: Drug: Lopinavir/ritonavir

INTERVENTIONS:
Drug: Darunavir/ritonavir — Darunavir/ritonavir 800/100 mg once daily
  Other Names: N/P
  Arms: Darunavir/ritonavir
Drug: Lopinavir/ritonavir — Lopinavir/ritonavir 400/100 mg twice daily
  Other Names: N/P
  Arms: Lopinavir/ritonavir

SUMMARY:
The purpose of this study is to determine the non-inferiority in the efficacy of DRV/r (900/100 mg) monotherapy at 48 weeks versus LPV/r (400/100 mg) as simplification strategy in subjects with sustained viral suppression on stable PI or NNRTI-antiretroviral regimens.

DETAILED DESCRIPTION:
The pillar of the current standard of care for highly active antiretroviral therapies (HAART) is the use of two nucleoside reverse transcriptase inhibitors (NRTIs).1 However, these agents can inhibit the mitochondrial DNA polymerase gamma, causing mitochondrial dysfunction, which, in turn, may cause NRTI-related adverse events such as peripheral neuropathy, pancreatitis, liver disturbances, lipid profile abnormalities or lipoatrophy.2 As a result, strategies aimed to avoid the long term exposure to NRTIs and their toxicities are desirable for the management of HIV-infected patients.

Monotherapy with protease inhibitors (PIs) as a simplification approach therapy after an induction period with conventional antiretroviral treatment, appears to be of great utility for minimizing mitochondrial toxicity because of NRTIs. This approach may also increase patient adherence, reduce costs and preserve future treatment options. However, concerns remain regarding compartmental HIV replication due to limited drug penetration into the central nervous system, risk factors associated with monotherapy failure as well as the extrapolation of results obtained in clinical trial settings to routine clinical practice, are still not well known.

In this regard, there are reports that have suggested that lopinavir/ritonavir (LPV/r) monotherapy may be an effective therapeutic option for treatment of HIV-1 infection in antiretroviral-naïve patients. 5,6 Moreover, some studies report that despite LPV/r allows CSF concentrations lower than plasma, its concentrations exceed levels that suppress wild-type HIV replication.7,8,9 However other authors have reported that LPV/r monotherapy results in suboptimal HIV suppression in the CSF compartment in approximately 10% of cases.10

Darunavir is the last PI with activity against wild-type and PI-resistant HIV. In ARTEMIS trial, DRV/r at doses of 800/100 mg once daily have demonstrated that it is non inferior and statistically superior than LPV/r and it is an effective treatment option for antiretroviral (ARV)-naïve patients. In this study, patients receiving once-daily DRV/r achieved high durable virologic response rates, which were comparable in patients with less favourable baseline characteristics or suboptimal adherence. In addition, they had a low discontinuation rate due to virologic failure or adverse events or both, did not develop protease inhibitor resistance upon failure, and had suitable drug exposure. 11,12

All these benefits, coupled with the higher genetic barrier, its favourable safety and plasmatic pharmacokinetic profile of DRV/r, suggest that DRV/r has the potential to be an excellent option for monotherapy simplification strategies.

The investigators propose a prospective and randomised clinical trial that compares the efficacy, safety and tolerability of DRV/r 900/100 mg monotherapy once daily versus LPV/r 400/100 monotherapy twice daily as simplification strategy in HIV-infected patients with stable NNRTI or PI-based antiretroviral regimen and sustained viral suppression.

Aside to the main goal of this project, the investigators are going to make use of the samples obtained from the CSF at 48 weeks of follow-up (as representative of the viruses replicating in the central nervous system) and genital tract and plasma at the different time points. The investigators will compare the sequence population of those organs from the different patients in order to state if viruses not found in plasma at one time point but found in reservoirs can be found in blood when the infection advance.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected adults (=/+18 years old).
* Patients having a diagnosis of HIV infection, on stable HAART including:

  2 NRTI/NtRTIs plus one of the following : 1 PI/ritonavir (lopinavir/ritonavir, atazanavir/ritonavir, fosamprenavir /ritonavir, tipranavir/ritonavir, darunavir/ritonavir) or ATV/unboosted (in a regimen without tenofovir) 1 NNRTI (nevirapine or efavirenz), raltegravir or maraviroc
* Undetectable plasma HIV-1 RNA (VL < 50 copies/mL) while on HAART during at least 3 month prior to switching.
* Nadir CD4 cell count > 100 cells/mm3.
* Absence of major PI-resistance mutations in HIV-protease (IAS 2008).20 Good treatment adherence.
* Voluntary written informed consent.
* Patients and physician's preference to change the current HAART regimen for reasons of simplification and/or toxicity.

Exclusion Criteria:

* History of virological failure to a previous antiretroviral protease-containing regimens.
* History of virological failure defined as two consecutive plasma HIV-1 RNA > 50 copies/mL while on current antiretroviral therapy
* Acute infections or uncontrolled chronic infection in the 2 months previous to the inclusion or physical examination that, in the investigator's opinion, would compromise the patient's safety or outcome of the study
* Breastfeeding, pregnancy or fertile women willing to be pregnant.
* Patients co-infected with hepatitis B.
* Concomitant use of any drug with potential drug-drug interaction with DRV/r or LPV/r at study entry.
* Therapies including interferon, interleukin-2, cytotoxic chemotherapy or immunosuppressors at study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Plasmatic HIV-1 Viral load | week 48

SECONDARY OUTCOMES:
CD4 cell count | baseline, weeks 12, 24, 36, 48
Changes in liver enzymes (aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma GT, alkaline phosphatase) | baseline, weeks 12, 24, 36, 48
Changes in total bilirubin | baseline, weeks 12, 24, 36, 48
Changes in lipid parameters (total, HDL-, LDL-, cholesterol, triglycerides) | baseline, weeks 12, 24, 36, 48
Administration of lipid-lowering drugs throughout the study (new administrations or the withdrawal of previous lipid-lowering drugs) | baseline, weeks 4, 12, 24, 36, 48.
Adverse events | weeks 4, 12, 24, 36, 48.
CSF and genital tract HIV-1 viral load | baseline, weeks 24, 48
Plasmatic, CSF and genital tract trough-DRV and LPV concentration | weeks 12, 24, 48
Resistance mutations in case of confirmed virological failure (plasmatic, CSF and genital tract) | baseline, weeks 4, 12, 24, 36, 48.
Neurocognitives changes | baseline, week 48
Time to virological failure, defined as an increase in HIV RNA >50 copies in 2 determinations within 1 month. The first date with VL > 50 will be used to calculate time to virological failure. | weeks 4, 12, 24, 36, 48.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Germans Trias i Pujol Hospital, Badalona, Barcelona
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands